CLINICAL TRIAL: NCT04184648
Title: Clinical Study on Comparative Diagnostic Criteria of Bronchopulmonary Dysplasia in Premature Infants
Brief Title: Comparison of Classification Standards of BPD in Premature Infants
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Wang Jianhui (Other)
Responsible Party: Sponsor-Investigator, Wang Jianhui, principal investigator, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Other Study IDs: 00020191112
Record Dates: First submitted 2019-11-29; First posted 2019-12-03 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary Dysplasia; high-flow nasal cannula; noninvasive ventilation; Ventilation mode; premature infant
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- There was no adverse systems outcome after PMA36 weeks: Premature infants at PMA36 weeks did not show the following conditions (1) before follow-up tracheotomy; (2) the duration of hospital stay exceeds 50 weeks of PMA; (3) continuous or intermittent use of oxygen and respiratory support for more than 12 months after birth; (4) readmission ≥2 times due to respiratory factors within 12 months. (5) death
  Interventions: Other: no interventions
- Death or adverse respiratory outcome after 36 weeks of pma: Premature infants at PMA36 weeks presented the following conditions (1) before tracheotomy during follow-up; (2) the duration of hospital stay exceeds 50 weeks of PMA; (3) continuous or intermittent use of oxygen and respiratory support for more than 12 months after birth; (4) readmission ≥2 times due to respiratory factors within 12 months. (5) death
  Interventions: Other: no interventions

INTERVENTIONS:
Other: no interventions — no intervention

SUMMARY:
Bronchopulmonary dysplasia of premature infants is a common respiratory disease in premature infants. Long-term complications such as recurrent respiratory infection and abnormal lung function may occur in the survivors, and may increase the risk of dysplasia of the nervous system. In the past 30 years, although the monitoring and treatment technology of premature infants has been significantly improved, the incidence of BPD still shows no downward trend, and effective treatment and prevention methods for BPD are still lacking. The progress of clinical research on BPD is slow, one of the important reasons is that the definition of BPD is still not consistent, and its diagnostic and grading standards lack objectivity. To summarize the development of diagnostic criteria for BPD in the past 30 years, there are still the following disadvantages. 1. 2. In the above study, all proposed alternative BPD classification standards did not completely separate HFNC and NIV. In view of this, this study separated HFNC and other NIV to form a new revised BPD classification standard. On this basis, a nested case-control study was conducted to compare the differences between the newly proposed classification standards and NICHD standards in 2001, Rosemary standards in 2018 and Jensen standards in predicting long-term respiratory outcomes and other systemic complications in premature infants, so as to provide a standard for more accurate diagnosis and evaluation of BPD in premature infants.

ELIGIBILITY:
Inclusion Criteria:

* premature infants whose gestational age is less than 32 weeks;
* hospital stay ≥14 days;
* complete clinical medical records, including effective follow-up information

Exclusion Criteria:

* congenital heart and lung malformation and specific chromosomal diseases;
* children abandon treatment halfway;
* death of children due to factors other than respiratory system.

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All premature infants whose gestational age is less than 32 weeks admitted to the neonatal department of children's hospital of chongqing medical university from January 2018 to May 2019 were in line with this study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-20 (Estimated); Study Completion 2022-06-29 (Estimated)

PRIMARY OUTCOMES:
mortality | through study completion, an average of 12 months
  the proportion of dead BPD infants against the total BPD infants in corresponding group
serious respiratory mobidities | up to 18 months after birth
  occurence of at least one of the following:(1) before follow-up tracheotomy; (2) the duration of hospital stay exceeds 50 weeks of PMA; (3) continuous or intermittent use of oxygen and respiratory support for more than 12 months after birth; (4) readmission ≥2 times due to respiratory factors within 12 months.
Follow-up of neurological development | up to 18 months after birth
  occurence of at least one of the following:(1) TIMP score ≤ reference P25, or bayley-3 cognitive or motor score < 85; (2) abnormal hearing screening or BAEP for two times; (3) abnormal ROP screening

SECONDARY OUTCOMES:
Length of first hospital stay | up to PMA 36 weeks
  days
days of oxygen supplement | up to 18 months after birth
  days during which the infants were given oxygen supplement
Pulmonary imaging findings | up to PMA 36 weeks
  result of X-ray
Oxygen way | up to 18 months after birth
  Changes in assisted ventilation
physical development outcome | up to 18 months after birth
  including length, weight, head circumference

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shi, M.D, Study Director — Children's Hospital of Chongqing Medical University
Locations (1):
- Children's hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Result] Iyengar A, Davis JM. Drug therapy for the prevention and treatment of bronchopulmonary dysplasia. Front Pharmacol. 2015 Feb 16;6:12. doi: 10.3389/fphar.2015.00012. eCollection 2015. PMID 25762933
- [Result] Shennan AT, Dunn MS, Ohlsson A, Lennox K, Hoskins EM. Abnormal pulmonary outcomes in premature infants: prediction from oxygen requirement in the neonatal period. Pediatrics. 1988 Oct;82(4):527-32. PMID 3174313
- [Result] Poindexter BB, Feng R, Schmidt B, Aschner JL, Ballard RA, Hamvas A, Reynolds AM, Shaw PA, Jobe AH; Prematurity and Respiratory Outcomes Program. Comparisons and Limitations of Current Definitions of Bronchopulmonary Dysplasia for the Prematurity and Respiratory Outcomes Program. Ann Am Thorac Soc. 2015 Dec;12(12):1822-30. doi: 10.1513/AnnalsATS.201504-218OC. PMID 26397992
- [Result] Meyer S, Franz AR, Bay J, Gortner L; NeoVitaA Study Group. Developing a better and practical definition of bronchopulmonary dysplasia. Acta Paediatr. 2017 May;106(5):842. doi: 10.1111/apa.13783. Epub 2017 Mar 13. No abstract available. PMID 28196293
- [Result] Higano NS, Spielberg DR, Fleck RJ, Schapiro AH, Walkup LL, Hahn AD, Tkach JA, Kingma PS, Merhar SL, Fain SB, Woods JC. Neonatal Pulmonary Magnetic Resonance Imaging of Bronchopulmonary Dysplasia Predicts Short-Term Clinical Outcomes. Am J Respir Crit Care Med. 2018 Nov 15;198(10):1302-1311. doi: 10.1164/rccm.201711-2287OC. PMID 29790784
- [Result] Higgins RD, Jobe AH, Koso-Thomas M, Bancalari E, Viscardi RM, Hartert TV, Ryan RM, Kallapur SG, Steinhorn RH, Konduri GG, Davis SD, Thebaud B, Clyman RI, Collaco JM, Martin CR, Woods JC, Finer NN, Raju TNK. Bronchopulmonary Dysplasia: Executive Summary of a Workshop. J Pediatr. 2018 Jun;197:300-308. doi: 10.1016/j.jpeds.2018.01.043. Epub 2018 Mar 16. No abstract available. PMID 29551318
- [Result] Jensen EA, Dysart K, Gantz MG, McDonald S, Bamat NA, Keszler M, Kirpalani H, Laughon MM, Poindexter BB, Duncan AF, Yoder BA, Eichenwald EC, DeMauro SB. The Diagnosis of Bronchopulmonary Dysplasia in Very Preterm Infants. An Evidence-based Approach. Am J Respir Crit Care Med. 2019 Sep 15;200(6):751-759. doi: 10.1164/rccm.201812-2348OC. PMID 30995069
- [Result] Kotecha SJ, Adappa R, Gupta N, Watkins WJ, Kotecha S, Chakraborty M. Safety and Efficacy of High-Flow Nasal Cannula Therapy in Preterm Infants: A Meta-analysis. Pediatrics. 2015 Sep;136(3):542-53. doi: 10.1542/peds.2015-0738. Epub 2015 Aug 17. PMID 26283781
- [Result] Hong H, Li XX, Li J, Zhang ZQ. High-flow nasal cannula versus nasal continuous positive airway pressure for respiratory support in preterm infants: a meta-analysis of randomized controlled trials. J Matern Fetal Neonatal Med. 2021 Jan;34(2):259-266. doi: 10.1080/14767058.2019.1606193. Epub 2019 Apr 24. PMID 30966839
- [Result] Kadivar M Md, Mosayebi Z Md, Razi N Md, Nariman S Md, Sangsari R Md. High Flow Nasal Cannulae versus Nasal Continuous Positive Airway Pressure in Neonates with Respiratory Distress Syndrome Managed with INSURE Method: A Randomized Clinical Trial. Iran J Med Sci. 2016 Nov;41(6):494-500. PMID 27853329